CLINICAL TRIAL: NCT02704481
Title: Non-surgical Alternatives to Treatment of Failed Medical Abortion: A Randomized Controlled Double-blind Trial
Brief Title: Non-surgical Alternatives to Treatment of Failed Medical Abortion
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding mechanism compromised
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1035
Record Dates: First submitted 2016-03-02; First posted 2016-03-10 (Estimated); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Abortion Failure
Keywords: mifepristone; misoprostol; medical abortion
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mifepristone-misoprostol (Experimental): Women randomized to receive 200 mg mifepristone to take on Day 1, 800 mcg buccal misoprostol to take 24-48 hours after later, and four placebo misoprostol pills to take a further 3-12 hours later.
  Interventions: Drug: Mifepristone; Drug: Misoprostol; Drug: Placebo misoprostol
- Misoprostol-misoprostol (Experimental): Women randomized to receive a placebo mifepristone pill to take on Day 1 and two doses of 800 mcg buccal misoprostol, the first of which should be taken 24-48 hours after the placebo and the second of which should be taken 3-12 hours after the first misoprostol dose.
  Interventions: Drug: Misoprostol; Drug: Placebo mifepristone

INTERVENTIONS:
Drug: Mifepristone — 200mg oral mifepristone
  Other Names: Mifeprex
  Arms: Mifepristone-misoprostol
Drug: Misoprostol — 800mcg buccal misoprostol
  Other Names: Cytotec
Drug: Placebo mifepristone — Matching placebo pill of 200mg mifepristone
  Arms: Misoprostol-misoprostol
Drug: Placebo misoprostol — Matching placebo pills of 800mcg misoprostol
  Arms: Mifepristone-misoprostol

SUMMARY:
The primary outcome of this study is to compare the effectiveness of a second complete course of 200 mg mifepristone and 800 mcg misoprostol for ongoing pregnancy following mifepristone-misoprostol medical abortion.

DETAILED DESCRIPTION:
This is a multi-site double-blind, randomized controlled trial to assess treatment with a repeat mifepristone-misoprostol regimen and with a two-dose misoprostol-alone regimen in women who are diagnosed with ongoing pregnancy ≤77 days gestational age at 1-week follow-up after medical abortion. The sample will be stratified in two cohorts: women with ongoing pregnancies <= 56 days of gestation and women with ongoing pregnancies 57-77 days of gestation. Eligible women who agree to participate in the study will be randomly assigned to either Group 1 for treatment with 200 mg mifepristone followed in 24-48 hours by 800 mcg buccal misoprostol, followed by 4 misoprostol placebo pills 3-12 hours later, or to Group 2 for treatment with one mifepristone placebo pill, followed by 800 mcg buccal misoprostol 24-48 hours later and another 800 mcg dose repeated in 3-12 hours.

The study will also assess the acceptability of additional medication for ongoing pregnancy following an initial course of mifepristone-misoprostol medical abortion.

ELIGIBILITY:
Inclusion Criteria:

* Have ultrasound evidence of an ongoing pregnancy (embryo with cardiac activity) <= 77 days gestational age at follow-up after using a mifepristone-misoprostol regimen for termination of pregnancy
* Agree to comply with study procedures
* Able to consent to study participation

Exclusion Criteria:

* Have an ongoing pregnancy but did not take an initial course of mifepristone and misoprostol at the study site
* Are < 18 years old in US and Canadian sites
* Present with other medical abortion outcomes including persistent non-viable pregnancies or empty sac
* Are unable to provide contact information for follow-up purposes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
The proportion of women in each study group, by gestational age cohort, who have a successful abortion without recourse to surgical intervention for any reason. | One week after taking first study medication

SECONDARY OUTCOMES:
The proportion of women in each arm by gestational age cohort with resolved ongoing pregnancies following study treatment, regardless of surgical intervention | One week after taking first study medication
The proportion of women who found medical treatment to be an acceptable method to treat ongoing pregnancy, as measured by a follow up questionnaire | One week after taking first study medication

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Dzuba, MHS, Principal Investigator — Gynuity Health Projects; Tara Shochet, PhD, MPH, Principal Investigator — Gynuity Health Projects
Locations (14):
- United States (14):
  - Planned Parenthood of Northern California, Concord, California
  - Planned Parenthood of the Pacific Southwest, San Diego, California
  - Planned Parenthood of the Rocky Mountains, Denver, Colorado
  - Presidential Women's Center, West Palm Beach, Florida
  - Planned Parenthood of Illinois, Chicago, Illinois
  - Family Planning Associates Medical Group, Ltd., Chicago, Illinois
  - Planned Parenthood of the Heartland, Des Moines, Iowa
  - Emma Goldman Clinic, Iowa City, Iowa
  - Planned Parenthood of Northern New England, Topsham, Maine
  - Planned Parenthood League of Massachusetts, Boston, Massachusetts
  - Planned Parenthood of Mid and South Michigan, Ann Arbor, Michigan
  - Northland Family Planning Clinic Inc., Westland, Michigan
  - Planned Parenthood of Central and Greater Northern New Jersey, Morristown, New Jersey
  - Montefiore Family Health Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No